CLINICAL TRIAL: NCT03632993
Title: A Phase 2A, Open-Label Study Evaluating the Safety and Different Injection Techniques of CCH for the Treatment of Edematous Fibrosclerotic Panniculopathy (EFP)
Brief Title: Injection Techniques of Collagenase Clostridium Histolyticum (CCH) for the Treatment of EFP (Cellulite)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EN3835-209
Record Dates: First submitted 2018-07-05; First posted 2018-08-16 (Actual); Results first posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Edematous Skin
Keywords: Edematous Fibrosclerotic Panniculopathy; Cellulite; Collagenase Clostridium Histolyticum
MeSH Terms: conditions — Cellulite | interventions — Microbial Collagenase

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment I: CCH Shallow Injection, 3 Aliquots (Active Comparator): In Treatment I, CCH will be injected subcutaneously while the participant lies in a prone position. Each injection will consist of a single skin injection of study drug administered as three 0.1 milliliters (mL) aliquots (for a total injection volume of 0.3 mL).
  During each treatment visit, 8 syringes (4 syringes per treatment area) will be prepared for dosing. Each syringe will contain 0.9 mL of CCH (3 injections in each syringe). Dose per participant per treatment visit = up to 1.68 milligrams (mg) of CCH (0.84 mg in each treatment area).
  Interventions: Drug: collagenase clostridium histolyticum (CCH)
- Treatment II: CCH Shallow Injection, 1 Aliquot (Active Comparator): In Treatment II, CCH will be injected subcutaneously while the participant is in a prone position. Each injection will consist of a single skin injection of study drug administered as a single shallow injection of a 0.3 mL aliquot.
  During each treatment visit, 8 syringes (4 syringes per treatment area) will be prepared for dosing. Each syringe will contain 0.9 mL of CCH (3 injections in each syringe). Dose per participant per treatment visit = up to 1.68 mg of CCH (0.84 mg in each treatment area).
  Interventions: Drug: collagenase clostridium histolyticum (CCH)
- Treatment III: CCH Deep Injection, 1 Aliquot (Active Comparator): In Treatment III, CCH will be injected subcutaneously while the participant is in a prone position. Each injection will consist of a single skin injection of study drug administered as a single deep injection of a 0.3 mL study drug aliquot.
  During each treatment visit, 8 syringes (4 syringes per treatment area) will be prepared for dosing. Each syringe will contain 0.9 mL of CCH (3 injections in each syringe). Dose per participant per treatment visit = up to 1.68 mg of CCH (0.84 mg in each treatment area).
  Interventions: Drug: collagenase clostridium histolyticum (CCH)
- Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Active Comparator): In Treatment IV, CCH will be injected subcutaneously while the participant lies in a prone position. Each injection will consist of a single skin injection of study drug administered as five 0.3 mL (for a total injection volume of 1.5 mL).
  During each treatment visit, 24 syringes (12 syringes per treatment area) will be prepared for dosing. Each syringe will contain 1.5 mL of CCH (5 aliquots of 0.3 mL, for each injection, in each syringe). Dose per participant per treatment visit = up to 1.68 mg of CCH (0.84 mg in each treatment area).
  Interventions: Drug: collagenase clostridium histolyticum (CCH)
- Treatment V: CCH Shallow Injections, 4 Aliquots (Active Comparator): In Treatment V, CCH will be injected subcutaneously while the participant lies in a prone position. Each injection will receive a single skin injection of study drug administered as four 0.3 mL aliquots (for a total injection volume of 1.2 mL).
  During each treatment visit, 24 syringes (12 syringes per treatment area) will be prepared for dosing. Each syringe will contain 1.2 mL of CCH (4 aliquots of 0.3 mL each). Dose per participant per treatment visit = up to 1.68 mg of CCH (0.84 mg in each treatment area).
  Interventions: Drug: collagenase clostridium histolyticum (CCH)

INTERVENTIONS:
Drug: collagenase clostridium histolyticum (CCH) — Endo Pharmaceuticals Inc. (Endo) is developing collagenase clostridium histolyticum (CCH) for the treatment of EFP. Because CCH is a proteinase that can hydrolyze the triple-helical region of collagen under physiological conditions, CCH has the potential to be effective in lysing sub-dermal collagen, such as those observed in the dermal septa, which are the underlying cause of the skin dimpling in women with Edematous Fibrosclerotic Panniculopathy (EFP). CCH targets the collagenase structural matrix (for example, dermal septa) at the site of injection and does not require systemic exposure to be effective.

SUMMARY:
The study will evaluate the safety and effectiveness of different injection techniques of Collagenase Clostridium Histolyticum (CCH) for the treatment of adult women with mild, moderate or severe Edematous Fibrosclerotic Panniculopathy (commonly known as Cellulite).

ELIGIBILITY:
Inclusion Criteria:

No participant will be assigned to treatment until all eligibility criteria have been satisfied. To qualify for the study a participant must:

1. Be able to provide voluntary written informed consent prior to the initiation of any study specific procedures per the policy of the governing Institutional Review Board (IRB)/Independent Ethics Committee (IEC).
2. Be female and at least 18 years of age at the time of consent.
3. Have evidence of cellulite in 2 bilateral treatment areas (defined as right and left buttocks or right and left posterolateral thighs) as assessed by the Investigator at the Screening visit, and fulfills the following requirements:

   1. has a score of 2 (mild), 3 (moderate) or 4 (severe) as reported by the Investigator (CR-PCSS) in 2 treatment areas (two thighs or two buttocks) at the Screening Visit.
   2. has at least 2 dimples from each treatment area that:

      * are isolated and separated by at least 5 centimeters (cm) from any other dimples.
      * score 2 or 3 on the Hexsel depression scale.
      * have dimple width: length ratio ≥ 0.5.
4. Be willing to apply sunscreen to the dosing areas before each exposure to the sun while participating in the study (that is, screening through end of study).
5. Be judged to be in good health, based upon the results of a medical history, physical examination, and laboratory profile at screening.
6. Have a negative serum pregnancy test at the Screening Visit and negative urine pregnancy at Day 1 (before injection of study drug), be using an effective contraception method (for example, abstinence, intrauterine device, hormonal [estrogen/progestin] contraceptives, or double barrier control) for at least 1 menstrual cycle prior to study enrollment and through Day 71; or be menopausal defined as at least 12 months of amenorrhea in the absence of other biological or physiological causes (as determined by the Investigator), or be post-menopausal for at least 1 year, or be surgically sterile (hysterectomy, bilateral oophorectomy, bilateral tubal ligation).
7. Be willing and able to comply with all protocol required study visits and assessments.

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from the study:

1. Is pregnant or is intending to become pregnant during the study.
2. Is presently nursing/breastfeeding or providing breast milk.
3. Has any of the following systemic conditions:

   1. Coagulation disorder.
   2. Evidence or history of malignancy (other than excised basal-cell carcinoma) unless there has been no recurrence in at least 5 years.
   3. History of keloidal scarring or abnormal wound healing.
   4. Concurrent diseases or conditions that might interfere with the conduct of the study, confound the interpretation of the study results, or endanger the participant's well-being.
   5. Evidence of clinically significant abnormalities on physical examination, vital signs, electrocardiogram (ECG), or clinical laboratory values.
4. Has any of the following local conditions in the areas to be treated:

   1. History of lower extremity thrombosis or post-thrombosis syndrome.
   2. Vascular disorder (for example, varicose veins, telangiectasia).
   3. Inflammation or active infection.
   4. Severe skin laxity, flaccidity, and/or sagging.
   5. Active cutaneous alteration including rash, eczema, psoriasis, or skin cancer.
5. Has a tattoo located within 2 cm of the site of injection.
6. Requires anticoagulant or antiplatelet medication during the study or has received anticoagulant or antiplatelet medication (except for ≤ 150 mg aspirin daily) within 7 days before injection of study drug.
7. Has used any of the following for the treatment of EFP on the area to be treated within the timelines identified below or intends to use any of the following at any time during the course of the study:

   1. Liposuction within the treatment areas during the 12-month period before injection of study drug.
   2. Injections (for example, mesotherapy); radiofrequency device treatments; laser treatment; or surgery (including subcision and/or powered subcision) within the treatment areas during the 12-month period before injection of study drug.
   3. Any investigational treatment for EFP/cellulite on treatment areas during the 12-month period before the injection of study drug.
   4. Endermologie® or similar treatments within the treatment areas during the 6-month period before injection of study drug.
   5. Massage therapy within the treatment areas during the 3-month period before injection of study drug.
   6. Creams (for example, Celluvera™, TriLastin®) to prevent or mitigate EFP within the treatment areas during the 2-week period before injection of study drug.
8. Has received an investigational drug or treatment within 30 days before injection of study drug.
9. Has a known systemic allergy to collagenase or any other excipient of study drug.
10. Has a history of drug or alcohol abuse.
11. Intends to initiate an intensive sport or exercise program during the study.
12. Intends to initiate a weight reduction program during the study.
13. Intends to use tanning spray or tanning booths during the study.
14. Has previously received any collagenase treatments (for example, Santyl® ointment and/or XIAFLEX/XIAPEX®).
15. Was a participant in a previous cellulite clinical trial of EN3835: AUX-CC-830, AUX-CC-831, EN3835-102, EN3835-104, EN3835-201, EN3835-202, EN3835-205, EN3835-302, or EN3835-303.
16. Any other condition(s) that, in the Investigator's opinion, might indicate the participant is unsuitable for the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 64 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Omburo, Study Director — Endo Pharmaceuticals
Locations (5):
- United States (5):
  - Endo Clinical Trial Site #1, Coral Gables, Florida
  - Endo Clinical Trial Site #5, Miami, Florida
  - Endo Clinical Trial Site #2, New York, New York
  - Endo Clinical Trial Site #4, New York, New York
  - Endo Clinical Trial Site #3, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants in each treatment region (buttocks or thighs) were assigned to 1 of 5 injection technique treatment arms. No participants were treated in both the buttocks and the thighs.
Units Other Than Participants: buttocks or thighs
Groups:
- Treatment I: CCH Shallow Injection, 3 Aliquots (Buttocks): In Treatment I, each injection consisted of a single skin injection of study drug administered as a shallow injection of three 0.1 milliliters (mL) aliquots (for a total injection volume of 0.3 mL).
  Each participant received 24 injections for a total dose of 1.68 mg of CCH (0.84 mg per treatment region) at each treatment visit.
- Treatment I: CCH Shallow Injection, 3 Aliquots (Thighs): In Treatment I, each injection consisted of a single skin injection of study drug administered as a shallow injection of three 0.1 mL aliquots (for a total injection volume of 0.3 mL).
  Each participant received 24 injections for a total dose of 1.68 mg of CCH (0.84 mg per treatment region) at each treatment visit.
- Treatment II: CCH Shallow Injection, 1 Aliquot (Buttocks); Treatment II: CCH Shallow Injection, 1 Aliquot (Thighs): In Treatment II, each injection consisted of a single skin injection of study drug administered as a single shallow injection of a 0.3 mL aliquot.
  Each participant received 24 injections for a total dose of 1.68 mg of CCH (0.84 mg per treatment region) at each treatment visit.
- Treatment III: CCH Deep Injection, 1 Aliquot (Buttocks); Treatment III: CCH Deep Injection, 1 Aliquot (Thighs): In Treatment III, each injection consisted of a single skin injection of study drug administered as a single deep injection of a 0.3 mL study drug aliquot.
  Each participant received 24 injections for a total dose of 1.68 mg of CCH (0.84 mg per treatment region) at each treatment visit.
- Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Buttocks); Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Thighs): In Treatment IV, each injection consisted of a single skin injection of study drug administered as five 0.3 mL aliquots (one deep and four shallow; total injection volume of 1.5 mL).
  Each participant received 24 injections for a total dose of 1.68 mg of CCH (0.84 mg per treatment region) at each treatment visit.
- Treatment V: CCH Shallow Injections, 4 Aliquots (Buttocks); Treatment V: CCH Shallow Injections, 4 Aliquots (Thighs): In Treatment V, each injection consisted of a single skin injection of study drug administered as a shallow injection of four 0.3 mL aliquots (for a total injection volume of 1.2 mL).
  Each participant received 24 injections for a total dose of 1.68 mg of CCH (0.84 mg per treatment region) at each treatment visit.
Period: Overall Study
Arm/Group | Treatment I: CCH Shallow Injection, 3 Aliquots (Buttocks) | Treatment I: CCH Shallow Injection, 3 Aliquots (Thighs) | Treatment II: CCH Shallow Injection, 1 Aliquot (Buttocks) | Treatment II: CCH Shallow Injection, 1 Aliquot (Thighs) | Treatment III: CCH Deep Injection, 1 Aliquot (Buttocks) | Treatment III: CCH Deep Injection, 1 Aliquot (Thighs) | Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Buttocks) | Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Thighs) | Treatment V: CCH Shallow Injections, 4 Aliquots (Buttocks) | Treatment V: CCH Shallow Injections, 4 Aliquots (Thighs)
Started | 7; 14 buttocks or thighs (Treated in both buttocks) | 6; 12 buttocks or thighs (Treated in both thighs) | 6; 12 buttocks or thighs (Treated in both buttocks) | 7; 14 buttocks or thighs | 6; 12 buttocks or thighs (Treated in both buttocks) | 6; 12 buttocks or thighs (Treated in both thighs) | 6; 12 buttocks or thighs | 7; 14 buttocks or thighs | 7; 14 buttocks or thighs | 6; 12 buttocks or thighs
Completed | 6; 12 buttocks or thighs | 5; 10 buttocks or thighs | 6; 12 buttocks or thighs | 7; 14 buttocks or thighs | 6; 12 buttocks or thighs | 4; 8 buttocks or thighs | 6; 12 buttocks or thighs | 5; 10 buttocks or thighs | 7; 14 buttocks or thighs | 5; 10 buttocks or thighs
Not Completed | 1; 2 buttocks or thighs | 1; 2 buttocks or thighs | 0; 0 buttocks or thighs | 0; 0 buttocks or thighs | 0; 0 buttocks or thighs | 2; 4 buttocks or thighs | 0; 0 buttocks or thighs | 2; 4 buttocks or thighs | 0; 0 buttocks or thighs | 1; 2 buttocks or thighs
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Non-compliance | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population includes all participants who had at least 1 injection of study drug.
Groups:
- Treatment I: CCH Shallow Injection, 3 Aliquots (Buttocks); Treatment I: CCH Shallow Injection, 3 Aliquots (Thighs): In Treatment I, each injection consisted of a single skin injection of study drug administered as a shallow injection of three 0.1 mL aliquots (for a total injection volume of 0.3 mL).
  Each participant received 24 injections for a total dose of 1.68 mg of CCH (0.84 mg per treatment region) at each treatment visit.
- Total: Total of all reporting groups
Arm/Group | Treatment I: CCH Shallow Injection, 3 Aliquots (Buttocks) | Treatment I: CCH Shallow Injection, 3 Aliquots (Thighs) | Treatment II: CCH Shallow Injection, 1 Aliquot (Buttocks) | Treatment II: CCH Shallow Injection, 1 Aliquot (Thighs) | Treatment III: CCH Deep Injection, 1 Aliquot (Buttocks) | Treatment III: CCH Deep Injection, 1 Aliquot (Thighs) | Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Buttocks) | Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Thighs) | Treatment V: CCH Shallow Injections, 4 Aliquots (Buttocks) | Treatment V: CCH Shallow Injections, 4 Aliquots (Thighs) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6 | 6 | 6 | 7 | 7 | 6 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (9.85) | 44.7 (8.19) | 43.3 (10.95) | 45.6 (9.55) | 48.7 (15.95) | 52.2 (13.04) | 51.5 (11.93) | 49.0 (12.75) | 48.4 (10.00) | 39.8 (10.26) | 47.3 (11.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 6 | 7 | 6 | 6 | 6 | 7 | 7 | 6 | 63
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 3 | 6 | 3 | 1 | 1 | 2 | 5 | 3 | 32
  Not Hispanic or Latino | 2 | 2 | 3 | 1 | 3 | 5 | 5 | 5 | 2 | 3 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 2 | 1 | 0 | 1 | 0 | 3 | 1 | 3 | 14
  White | 3 | 6 | 4 | 6 | 6 | 5 | 5 | 4 | 6 | 3 | 48
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 90.258 (30.2437) | 75.660 (15.2730) | 87.843 (23.6933) | 84.407 (20.2152) | 76.687 (13.3870) | 74.117 (13.9682) | 65.038 (17.0083) | 72.396 (15.6629) | 78.497 (12.0413) | 96.008 (14.9791) | 80.012 (19.0943)
Height [Mean (Standard Deviation); unit: cm] — Population: One participant did not have data collected for height.
  cm
    number analyzed (Participants) | 6 | 5 | 6 | 7 | 6 | 6 | 6 | 7 | 7 | 6 | 62
    (all) | 158.7 (3.67) | 162.2 (3.03) | 161.8 (2.14) | 164.4 (10.01) | 163.0 (6.90) | 162.3 (3.88) | 161.5 (8.96) | 167.4 (10.55) | 164.4 (8.96) | 165.2 (6.65) | 163.2 (7.18)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: One participant did not have data collected for BMI.
  kg/m^2
    number analyzed (Participants) | 6 | 5 | 6 | 7 | 6 | 6 | 6 | 7 | 7 | 6 | 62
    (all) | 35.92 (12.643) | 30.30 (6.387) | 33.65 (9.415) | 31.11 (6.277) | 29.13 (6.239) | 28.05 (4.669) | 24.78 (5.202) | 26.40 (7.330) | 29.01 (4.123) | 35.10 (3.929) | 30.27 (7.379)
Skin Category (Fitzpatrick Scale) [Count of Participants; unit: Participants]
  I (Pale White) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  II (Fair) | 1 | 2 | 1 | 0 | 2 | 1 | 1 | 2 | 2 | 0 | 12
  III (Darker White) | 0 | 2 | 0 | 0 | 2 | 3 | 3 | 0 | 1 | 0 | 11
  IV (Light Brown) | 2 | 2 | 3 | 6 | 2 | 1 | 1 | 0 | 3 | 3 | 23
  V (Brown) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 3 | 7
  VI (Dark Brown or Black) | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 9

OUTCOME MEASURES:

1. Primary Outcome: Aesthetic Appearance Improvement Likert Scores by Treatment Region at Day 22
Description: Aesthetic appearance improvement for each treatment area (buttocks or thighs) was assessed by a blinded central assessment, using a 5-point Likert scale with scores ranging from -1 to 3. Aesthetic improvement was scored as worse (-1), stayed the same (0), improved (1), much improved (2) and very much improved (3). The assessor evaluated the image at Day 22 in comparison with baseline and recorded the Likert score. Aesthetic appearance Likert scale scores were analyzed using linear mixed model with treatment arm, study visit, interaction of treatment arm and study visit as fixed effects. This model was fitted using the response for the average of left and right of treatment area (that is, average of left buttock and right buttock or average of left thigh and right thigh).
Time Frame: Day 22
Population: Evaluable Population includes all participants in the Safety Population who had completed screening procedures and at least 1 baseline assessment of aesthetic appearance improvement Likert scale rating at specified timepoint. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for the assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment I: CCH Shallow Injection, 3 Aliquots (Buttocks) | Treatment I: CCH Shallow Injection, 3 Aliquots (Thighs) | Treatment II: CCH Shallow Injection, 1 Aliquot (Buttocks) | Treatment II: CCH Shallow Injection, 1 Aliquot (Thighs) | Treatment III: CCH Deep Injection, 1 Aliquot (Buttocks) | Treatment III: CCH Deep Injection, 1 Aliquot (Thighs) | Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Buttocks) | Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Thighs) | Treatment V: CCH Shallow Injections, 4 Aliquots (Buttocks) | Treatment V: CCH Shallow Injections, 4 Aliquots (Thighs)
Number analyzed (Participants) | 6 | 5 | 6 | 7 | 6 | 5 | 6 | 6 | 7 | 5
score on a scale | 1.08 [0.51 to 1.65] | 1.10 [0.46 to 1.74] | 0.75 [0.18 to 1.32] | 0.50 [-0.04 to 1.04] | 0.67 [0.10 to 1.24] | 0.20 [-0.44 to 0.84] | 0.83 [0.26 to 1.40] | 0.67 [0.09 to 1.25] | 1.00 [0.47 to 1.53] | 1.10 [0.46 to 1.74]

2. Primary Outcome: Aesthetic Appearance Improvement Likert Scores by Treatment Region at Day 43
Description: Aesthetic appearance improvement for each treatment area (buttocks or thighs) was assessed by a blinded central assessment, using a 5-point Likert scale with scores ranging from -1 to 3. Aesthetic improvement was scored as worse (-1), stayed the same (0), improved (1), much improved (2) and very much improved (3). The assessor evaluated the image at Day 43 in comparison with baseline and recorded the Likert score. Aesthetic appearance Likert scale scores were analyzed using linear mixed model with treatment arm, study visit, interaction of treatment arm and study visit as fixed effects. This model was fitted using the response for the average of left and right of treatment area (that is, average of left buttock and right buttock or average of left thigh and right thigh).
Time Frame: Day 43
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment I: CCH Shallow Injection, 3 Aliquots (Buttocks) | Treatment I: CCH Shallow Injection, 3 Aliquots (Thighs) | Treatment II: CCH Shallow Injection, 1 Aliquot (Buttocks) | Treatment II: CCH Shallow Injection, 1 Aliquot (Thighs) | Treatment III: CCH Deep Injection, 1 Aliquot (Buttocks) | Treatment III: CCH Deep Injection, 1 Aliquot (Thighs) | Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Buttocks) | Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Thighs) | Treatment V: CCH Shallow Injections, 4 Aliquots (Buttocks) | Treatment V: CCH Shallow Injections, 4 Aliquots (Thighs)
Number analyzed (Participants) | 6 | 5 | 5 | 7 | 6 | 5 | 6 | 6 | 7 | 5
score on a scale | 0.75 [0.18 to 1.32] | 1.40 [0.76 to 2.04] | 1.10 [0.47 to 1.73] | 0.57 [0.03 to 1.11] | 1.00 [0.43 to 1.57] | -0.01 [-0.64 to 0.64] | 1.17 [0.60 to 1.74] | 0.42 [-0.16 to 1.00] | 1.21 [0.69 to 1.74] | 0.70 [0.06 to 1.34]

3. Primary Outcome: Aesthetic Appearance Improvement Likert Scores by Treatment Region at Day 71
Description: Aesthetic appearance improvement for each treatment area (buttocks or thighs) was assessed by a blinded central assessment, using a 5-point Likert scale with scores ranging from -1 to 3. Aesthetic improvement was scored as worse (-1), stayed the same (0), improved (1), much improved (2) and very much improved (3). The assessor evaluated the image at Day 71 in comparison with baseline and recorded the Likert score. Aesthetic appearance Likert scale scores were analyzed using linear mixed model with treatment arm, study visit, interaction of treatment arm and study visit as fixed effects. This model was fitted using the response for the average of left and right of treatment area (that is, average of left buttock and right buttock or average of left thigh and right thigh).
Time Frame: Day 71
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment I: CCH Shallow Injection, 3 Aliquots (Buttocks) | Treatment I: CCH Shallow Injection, 3 Aliquots (Thighs) | Treatment II: CCH Shallow Injection, 1 Aliquot (Buttocks) | Treatment II: CCH Shallow Injection, 1 Aliquot (Thighs) | Treatment III: CCH Deep Injection, 1 Aliquot (Buttocks) | Treatment III: CCH Deep Injection, 1 Aliquot (Thighs) | Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Buttocks) | Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Thighs) | Treatment V: CCH Shallow Injections, 4 Aliquots (Buttocks) | Treatment V: CCH Shallow Injections, 4 Aliquots (Thighs)
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6 | 4 | 6 | 5 | 7 | 5
score on a scale | 1.08 [0.51 to 1.65] | 0.92 [0.34 to 1.50] | 1.08 [0.51 to 1.65] | 0.43 [-0.11 to 0.97] | 1.00 [0.43 to 1.57] | 0.12 [-0.59 to 0.84] | 0.50 [-0.07 to 1.07] | 0.30 [-0.34 to 0.94] | 1.29 [0.76 to 1.81] | 0.60 [-0.04 to 1.24]

4. Primary Outcome: Change From Baseline in Dimple Depth Depression (Hexsel CSS [B]) by Treatment Region at Day 22
Description: Dimple depth depression for each treatment area was assessed by the Investigator using the Hexsel Cellulite Severity Scale (B). Dimple Depth Depression of Hexsel Cellulite Severity Scale (B) was assessed and graded as: no depression (0), superficial depressions (1), medium depth depressions (2) and deep depressions (3). A negative change in Hexsel CSS (B) from baseline indicated an improvement in depression depth. Change from Baseline in dimple depth depression of Hexsel Cellulite Severity Scale (B) was analyzed using linear mixed model with treatment arm, study visits, interaction of treatment arm and study visit as fixed effect. This model was fitted using the response for the average of left and right of treatment areas (that is, average of left buttock and right buttock; average of left thigh and right thigh)
Time Frame: Baseline, Day 22
Population: Evaluable Population includes all participants in the Safety Population who had completed screening procedures and at least 1 baseline assessment of aesthetic appearance Likert scale rating at specified timepoint. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for the assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment I: CCH Shallow Injection, 3 Aliquots (Buttocks) | Treatment I: CCH Shallow Injection, 3 Aliquots (Thighs) | Treatment II: CCH Shallow Injection, 1 Aliquot (Buttocks) | Treatment II: CCH Shallow Injection, 1 Aliquot (Thighs) | Treatment III: CCH Deep Injection, 1 Aliquot (Buttocks) | Treatment III: CCH Deep Injection, 1 Aliquot (Thighs) | Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Buttocks) | Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Thighs) | Treatment V: CCH Shallow Injections, 4 Aliquots (Buttocks) | Treatment V: CCH Shallow Injections, 4 Aliquots (Thighs)
Number analyzed (Participants) | 6 | 5 | 6 | 7 | 6 | 5 | 6 | 6 | 7 | 5
score on a scale | -0.83 [-1.28 to -0.39] | -0.30 [-0.84 to 0.24] | -0.17 [-0.61 to 0.28] | -0.43 [-0.89 to 0.03] | -0.17 [-0.61 to 0.28] | -0.20 [-0.74 to 0.34] | -0.83 [-1.28 to -0.39] | -0.67 [-1.16 to -0.17] | -0.14 [-0.56 to 0.27] | -0.20 [-0.74 to 0.34]

5. Primary Outcome: Change From Baseline in Dimple Depth Depression (Hexsel CSS [B]) by Treatment Region at Day 43
Description: as for outcome 4
Time Frame: Baseline, Day 43
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment I: CCH Shallow Injection, 3 Aliquots (Buttocks) | Treatment I: CCH Shallow Injection, 3 Aliquots (Thighs) | Treatment II: CCH Shallow Injection, 1 Aliquot (Buttocks) | Treatment II: CCH Shallow Injection, 1 Aliquot (Thighs) | Treatment III: CCH Deep Injection, 1 Aliquot (Buttocks) | Treatment III: CCH Deep Injection, 1 Aliquot (Thighs) | Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Buttocks) | Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Thighs) | Treatment V: CCH Shallow Injections, 4 Aliquots (Buttocks) | Treatment V: CCH Shallow Injections, 4 Aliquots (Thighs)
Number analyzed (Participants) | 6 | 5 | 5 | 7 | 6 | 5 | 6 | 6 | 7 | 5
score on a scale | -0.92 [-1.36 to -0.47] | -0.40 [-0.94 to 0.14] | -0.40 [-0.89 to 0.09] | -0.43 [-0.89 to 0.03] | -0.50 [-0.95 to -0.05] | -0.40 [-0.94 to 0.14] | -0.83 [-1.28 to -0.39] | -0.67 [-1.16 to -0.17] | -0.36 [-0.77 to 0.06] | -0.60 [-1.14 to -0.06]

6. Primary Outcome: Change From Baseline in Dimple Depth Depression (Hexsel CSS [B]) by Treatment Region at Day 71
Description: as for outcome 4
Time Frame: Baseline, Day 71
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment I: CCH Shallow Injection, 3 Aliquots (Buttocks) | Treatment I: CCH Shallow Injection, 3 Aliquots (Thighs) | Treatment II: CCH Shallow Injection, 1 Aliquot (Buttocks) | Treatment II: CCH Shallow Injection, 1 Aliquot (Thighs) | Treatment III: CCH Deep Injection, 1 Aliquot (Buttocks) | Treatment III: CCH Deep Injection, 1 Aliquot (Thighs) | Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Buttocks) | Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Thighs) | Treatment V: CCH Shallow Injections, 4 Aliquots (Buttocks) | Treatment V: CCH Shallow Injections, 4 Aliquots (Thighs)
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6 | 4 | 6 | 5 | 7 | 5
score on a scale | -1.17 [-1.61 to -0.72] | -0.33 [-0.83 to 0.16] | -0.08 [-0.53 to 0.36] | -0.29 [-0.74 to 0.17] | -0.67 [-1.11 to -0.22] | -0.75 [-1.36 to -0.14] | -0.83 [-1.28 to -0.39] | -1.40 [-1.94 to -0.86] | -0.36 [-0.77 to 0.06] | -0.80 [-1.34 to -0.26]

7. Secondary Outcome: Change From Baseline of Dimple Volume by Treatment Region
Description: For each treated buttock and thigh, 4 dimple parameters including the maximum length (largest straight line distance across the dimple), maximum width (largest straight line distance perpendicular to the maximum length measurement), surface are, and volume (between the base of the dimple and an interpolated surface) of the target dimple were assessed. A negative change from Day 1 indicated an improvement. Volume of Dimple from Day 1 pre-marking was analyzed using linear mixed model with treatment arm, study visit, interaction of treatment arm and study visit as fixed effects. This model was fitted using the measurement for the average of left and right of treatment areas (that is, average of left buttock posterior and right buttock posterior; average of left thigh lateral, left thigh oblique, left thigh posterior, right thigh lateral, right thigh oblique, and right thigh posterior).
Time Frame: Baseline, Day 22, Day 43, and Day 71
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: mm^3
Arm/Group | Treatment I: CCH Shallow Injection, 3 Aliquots (Buttocks) | Treatment I: CCH Shallow Injection, 3 Aliquots (Thighs) | Treatment II: CCH Shallow Injection, 1 Aliquot (Buttocks) | Treatment II: CCH Shallow Injection, 1 Aliquot (Thighs) | Treatment III: CCH Deep Injection, 1 Aliquot (Buttocks) | Treatment III: CCH Deep Injection, 1 Aliquot (Thighs) | Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Buttocks) | Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Thighs) | Treatment V: CCH Shallow Injections, 4 Aliquots (Buttocks) | Treatment V: CCH Shallow Injections, 4 Aliquots (Thighs)
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6 | 5 | 6 | 6 | 7 | 5
mm^3
  Day 22: number analyzed (Participants) | 6 | 5 | 6 | 7 | 6 | 5 | 6 | 6 | 7 | 5
  Day 22 | -0.01 [-0.04 to 0.01] | -0.02 [-0.07 to 0.02] | -0.001 [-0.03 to 0.02] | -0.04 [-0.08 to -0.0001] | -0.01 [-0.04 to 0.01] | 0.00 [-0.05 to 0.05] | -0.01 [-0.04 to 0.01] | -0.01 [-0.06 to 0.03] | -0.04 [-0.06 to -0.01] | -0.04 [-0.09 to 0.01]
  Day 43: number analyzed (Participants) | 6 | 5 | 5 | 7 | 6 | 5 | 6 | 6 | 7 | 5
  Day 43 | -0.02 [-0.05 to 0.00] | -0.03 [-0.08 to 0.02] | -0.02 [-0.05 to 0.00] | -0.04 [-0.08 to 0.00] | -0.01 [-0.04 to 0.01] | 0.01 [-0.04 to 0.06] | -0.01 [-0.04 to 0.01] | -0.02 [-0.07 to 0.02] | -0.04 [-0.07 to -0.02] | -0.06 [-0.11 to -0.01]
  Day 71: number analyzed (Participants) | 6 | 6 | 6 | 7 | 6 | 4 | 4 | 5 | 7 | 5
  Day 71 | -0.02 [-0.05 to 0.00] | -0.02 [-0.07 to 0.02] | -0.04 [-0.06 to -0.01] | -0.02 [-0.07 to 0.02] | -0.01 [-0.04 to 0.02] | 0.04 [-0.02 to 0.09] | -0.02 [-0.05 to 0.01] | -0.02 [-0.07 to 0.03] | -0.05 [-0.07 to -0.02] | -0.05 [-0.09 to 0.00]

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) through Day 71
Description: All (serious and nonserious) treatment-emergent adverse events, whether elicited or observed during study visits or spontaneously reported by the participant. Safety Population: All enrolled participants who received at least 1 injection of CCH.
Arm/Group | Treatment I: CCH Shallow Injection, 3 Aliquots (Buttocks) | Treatment I: CCH Shallow Injection, 3 Aliquots (Thighs) | Treatment II: CCH Shallow Injection, 1 Aliquot (Buttocks) | Treatment II: CCH Shallow Injection, 1 Aliquot (Thighs) | Treatment III: CCH Deep Injection, 1 Aliquot (Buttocks) | Treatment III: CCH Deep Injection, 1 Aliquot (Thighs) | Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Buttocks) | Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Thighs) | Treatment V: CCH Shallow Injections, 4 Aliquots (Buttocks) | Treatment V: CCH Shallow Injections, 4 Aliquots (Thighs)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 0/6 | 0/6 | 0/7 | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 0/6 | 0/6 | 1/7 | 1/7 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 4/6 | 7/7 | 6/6 | 6/6 | 6/6 | 7/7 | 7/7 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment I: CCH Shallow Injection, 3 Aliquots (Buttocks) (N=6) | Treatment I: CCH Shallow Injection, 3 Aliquots (Thighs) (N=6) | Treatment II: CCH Shallow Injection, 1 Aliquot (Buttocks) (N=6) | Treatment II: CCH Shallow Injection, 1 Aliquot (Thighs) (N=7) | Treatment III: CCH Deep Injection, 1 Aliquot (Buttocks) (N=6) | Treatment III: CCH Deep Injection, 1 Aliquot (Thighs) (N=6) | Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Buttocks) (N=6) | Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Thighs) (N=7) | Treatment V: CCH Shallow Injections, 4 Aliquots (Buttocks) (N=7) | Treatment V: CCH Shallow Injections, 4 Aliquots (Thighs) (N=6)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hospitalization (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment I: CCH Shallow Injection, 3 Aliquots (Buttocks) (N=6) | Treatment I: CCH Shallow Injection, 3 Aliquots (Thighs) (N=6) | Treatment II: CCH Shallow Injection, 1 Aliquot (Buttocks) (N=6) | Treatment II: CCH Shallow Injection, 1 Aliquot (Thighs) (N=7) | Treatment III: CCH Deep Injection, 1 Aliquot (Buttocks) (N=6) | Treatment III: CCH Deep Injection, 1 Aliquot (Thighs) (N=6) | Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Buttocks) (N=6) | Treatment IV: CCH Deep and Shallow Injections, 5 Aliquots (Thighs) (N=7) | Treatment V: CCH Shallow Injections, 4 Aliquots (Buttocks) (N=7) | Treatment V: CCH Shallow Injections, 4 Aliquots (Thighs) (N=6)
Injection site pain (General disorders) | 6 | 6 | 3 | 6 | 6 | 6 | 6 | 7 | 6 | 3
Injection site bruising (General disorders) | 5 | 4 | 4 | 7 | 6 | 6 | 3 | 3 | 5 | 6
Injection site nodule (General disorders) | 3 | 2 | 4 | 6 | 5 | 5 | 0 | 3 | 3 | 5
Injection site warmth (General disorders) | 2 | 4 | 2 | 3 | 2 | 0 | 1 | 1 | 2 | 2
Injection site pruritus (General disorders) | 3 | 3 | 1 | 3 | 2 | 0 | 2 | 1 | 2 | 0
Injection site haemorrhage (General disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 3 | 4 | 2 | 0
Injection site discolouration (General disorders) | 1 | 1 | 2 | 4 | 1 | 0 | 0 | 0 | 0 | 1
Injection site swelling (General disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 1
Injection site induration (General disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza-like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site mass (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Crystal urine present (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT03632993/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT03632993/SAP_001.pdf